CLINICAL TRIAL: NCT05596526
Title: Immunogenicity of the Recombinant Zoster Vaccine (Shingrix ®) in Multiple Sclerosis Patients Treated With Anti-CD20 Antibodies Compared to Controls- a Phase IV Monocentric Study
Brief Title: Immunogenicity of the Recombinant Zoster Vaccine in Multiple Sclerosis Patients
Acronym: MSHINGVAX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prof Patrice Lalive (Other)
Responsible Party: Sponsor-Investigator, Prof Patrice Lalive, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01255
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Shingles; Zoster
Keywords: RZV vaccine; Multiple Sclerosis; Immune response; Safety
MeSH Terms: conditions — Herpes Zoster; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS patients on anti-CD20 (Experimental): Participants aged 18 and above will receive two doses of the recombinant Zoster vaccine (Shingrix®)
  Interventions: Biological: recombinant zoster vaccine
- Healthy controls (Experimental): Healthy participants aged 50 to 59 will receive two doses of the recombinant Zoster vaccine (Shingrix®)
  Interventions: Biological: recombinant zoster vaccine

INTERVENTIONS:
Biological: recombinant zoster vaccine — Shingrix® vaccine will be administered in two vaccinations on Day0 and Day60
  Other Names: Shingrix®

SUMMARY:
The purpose of this study is to provide evidence as to whether RZV is immunogenic with an acceptable safety profile in Multiple Sclerosis patients on anti-CD20 treatment.

DETAILED DESCRIPTION:
In this monocentric study, we will assess the immunogenicity and safety of two doses of the adjuvanted recombinant Zoster vaccine (RZV, or Shingrix®) in Multiple sclerosis patients treated with anti-CD20 (ocrelizumab, group 1) compared to healthy controls (group 2).

Participants will receive Shingrix® on Day0 and Day60; immunological response will be assessed on Day 0, 1, Day 60, 61, Day90 and Day360.

Unsolicited Adverse events of special interest (AESI) will be collected throughout the study period; patients reported outcomes (PROs) will be declared for one week after each vaccination. Safety of MS patients will be monitored through EDSS scoring and MRI before and 1 month after vaccination (D90) and at day 180 and 360 (EDSS scoring only)

ELIGIBILITY:
Inclusion Criteria:

For MS patients:

* 18 years and above
* Diagnosed with relapsing MS according to McDonald Criteria (2017)
* Not already vaccinated by RZV and willing to be vaccinated with RZV.
* At least 1 year on anti-CD20 treatment: 2 initial infusions of Ocrelizumab 300 mg (2 weeks apart), one infusion of Ocrelizumab 600 mg 6 months apart, one infusion of Ocrelizumab 600 mg 12 months after initial infusions
* Informed consent as documented by signature

For healthy controls

* Aged 50 to 59
* Not already vaccinated by RZV and willing to be vaccinated with RZV
* Informed consent as documented by signature

Exclusion Criteria:

* Recent MS relapse in the 6 weeks preceding planned vaccination
* Ongoing signs of febrile or non-febrile infection at the time of vaccination
* Recent pregnancy with delivery in the six months preceding vaccination and/or planned pregnancy in the six months following RZV vaccination
* Immunosuppression from the following: HIV infection, current active systemic auto-immune disease (other than MS), current malignant neoplasm; primary immunodeficiency; recent solid or bone-marrow transplant or any transplant still requiring immunosuppressive therapy; conditions requiring medication with immunosuppressive drugs
* Having received a vaccine in the last month
* Having received a shingles vaccine within one year
* Presented with herpes zoster in the previous year
* Contra-indication to RZV
* Unable to provide informed consent or inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of glycoprotein E (gE)-specific total IgG | day 90
  gE-specific total Immunoglobulin(Ig)G titers is determined by gE-specific ELISA from sera samples

SECONDARY OUTCOMES:
Vaccine safety - AESI 7 days | 7 days
  Incidence adverse events of special interest (AESI) in the 7 days following each vaccination (reactogenicity) collected in a diary card
Vaccine safety - SAE 360 days | day 360
  Incidence of serious adverse events (SAE) throughout the study period
Vaccine safety -pIMDs | day 360
  Incidence of potential immune mediated disorders (pIMDs) throughout the study period
Vaccine safety-relapse in MS patients | day 90
  Incidence of relapse in MS patients during a follow-up of 3 months after the first dose (d90) compared to the year preceding vaccination with RZV
Vaccine immunogenicity - CD4+ T cells per million of T cells, measured at D90 | Day 90
  Mean of gE-specific CD4+ T cells expressing at least 2 activation markers (i.e. CD40 ligand, interferon-gamma, IL-2 or TNF-alpha) per million of T cells, measured at D90

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Lalive, Pr, Principal Investigator — University Hospitals of Geneva; Arnaud Didierlaurent, Pr, Study Director — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Shingrix vaccine information — https://www.ema.europa.eu/en/documents/product-information/shingrix-epar-product-information_en.pdf